CLINICAL TRIAL: NCT06814639
Title: "Index of Professional Governance" Tool: a Multicentric Validation and Measuring Professional Governance in an Italian Hospital Setting
Brief Title: The Aims of the Study Are to Translate the Index of Professional Governance (IPG 3.0) Into Italian and Validate It and to Assess the State of Professional Governance in an Italian Hospital (ISMETT)
Status: Not yet recruiting | Type: Observational
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Other Study IDs: IRRB/37/23
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Validation Study
Keywords: IPG tool; professional governance; translation; validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Professional Governance (PG) is a way to actualize better work environments and structural empowerment. PG has a history over many years in the healthcare industry and has been defined as multidimensional organizational characteristics that encompass the structure and processes through which professionals direct, control and regulate one another's goal-oriented efforts. Multiple studies over the years have shown that PG can lead to empowered personnel and quality of care delivered.

In many organizations, governance is primarily controlled by management. The responsibility for managing professional practice should, however, be shared by staff and leaders, and in order to empower staff, they should be engaged in identifying areas for improvement. In addition, evidence-based practice should be enabled by allocating sufficient time, research and access to evidence sources.

The participation element refers to who creates and participates in governance activities on different levels. Successful professional governance structures have been linked to a positive professional practice environment. An effective structure with true sharing of decision-making between management and personnel will also contribute to optimal patient outcomes.

To evaluate whether an organization's governance is empowering and professional, it must be measured. Thus, various instruments to measure nurses' participation in professional governance have been presented. The Index of Professional Nursing Governance (IPNG) has been used in more than 250 international healthcare organizations during the last 20 years to evaluate implementation of their management models.

Hess created the IPNG for measuring professional governance along a conceptual continuum from traditional, through shared to self-governance models. Hess has since continued to advance the questionnaire. At the same time, an extended tool was created with all professional figures involved, the so called "Index of Professional Governance" (IPG). Several revisions have been made over time up to the current version of the IPG 3.0 The IPG measures the governance of hospital-based professional, based on a model of governance derived from the literature, in 5 dimensions: personnel, information, resources, participation and practice. Those five dimensions are covered by 50 items. Respondents use a 5-point scale to identify the group that dominates certain areas of governance stated in the items, ranging from 'management/administration only' (1p), through 'equally shared by staff and management/administration' (3p) to 'staff only' (5p). The points for each dimension, and overall governance, are then organized together, analyzed and used to place the organization's governance on the continuum from traditional to self-governance.

Previously translated from its original language, English-American into Arabic, British, Finnish, French, German, Korean, Portuguese, it is structured in five dimensions: staff, information, resources, participation and practice. These 5 dimensions are analyzed in 50 items.

Aims of the study:

1. To translate the Index of Professional Governance (IPG 3.0) into Italian and validate it;
2. To assess the state of professional governance in an Italian hospital (ISMETT).

ELIGIBILITY:
Inclusion Criteria:

* 1 year of professional seniority
* possess adequate linguistic skills certified by passing an English test (prepared by the linguistic services of the promoting center).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Employees of 5 Italian hospital structures and representative of different professions (the administrative area, the nursing area, the area of the other health professions and the medical area).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-02-06 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Inter-rater agreement percentage in evaluating the conceptual equivalence of the italian translation of the IPG. | Feb-Mar 2025: Recruitment of evaluators and assessment of language proficiency. Apr-Sep 2025: Evaluation of the proposed and collection of evaluators' judgements and final approval of the translated items. Oct 2025: Final data analysis and study closure.